CLINICAL TRIAL: NCT05668091
Title: An Interventional Decentralized Phase 2, Randomized, Double-Blind, 2-Arm Study to Investigate the Efficacy and Safety of Orally Administered Nirmatrelvir/Ritonavir Compared with Placebo/Ritonavir in Participants with Long COVID
Brief Title: A Decentralized, Randomized Phase 2 Efficacy and Safety Study of Nirmatrelvir/Ritonavir in Adults with Long COVID.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harlan M Krumholz (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Harlan M Krumholz, Professor of Medicine, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000034086; CIICORE-01 (Other: Center for Infection and Immunity Center for Outcome Research and Evaluation)
Record Dates: First submitted 2022-12-24; First posted 2022-12-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Long COVID
Keywords: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir; Ritonavir; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nirmatrelvir / Ritonavir (Experimental): Participants receive nirmatrelvir plus ritonavir (Paxlovid) for 15 days. All 3 tablets (2 of nirmatrelvir and 1 of ritonavir) must be taken twice daily by mouth for 15 days.
  Interventions: Drug: Nirmatrelvir; Drug: Ritonavir
- Placebo / Ritonavir (Placebo Comparator): Participants receive placebo to match nirmatrelvir plus ritonavir for 15 days. The control formulation includes 2 placebo tablets and 1 ritonavir tablet.
  Interventions: Drug: Ritonavir; Drug: Placebo

INTERVENTIONS:
Drug: Nirmatrelvir — Two 150 mg tablets taken by mouth every 12 hours.
  Arms: Nirmatrelvir / Ritonavir
Drug: Ritonavir — One 100 mg capsule taken by mouth every 12 hours.
Drug: Placebo — Two tablets containing placebo matching nirmatrelvir taken by mouth every 12 hours.
  Other Names: sugar pill
  Arms: Placebo / Ritonavir

SUMMARY:
This decentralized trial is a Phase 2, 1:1 randomized, double-blind, superiority, placebo-controlled study in an anticipated 100 non-hospitalized highly symptomatic adult participants with long COVID. It seeks to determine the efficacy, safety, and tolerability of 15 days of Paxlovid (nirmatrelvir/ritonavir), an anti-viral agent, compared with placebo plus ritonavir. The hypothesis is that viral persistence contributes to long COVID in some patients and nirmatrelvir/ritonavir compared with placebo/ritonavir can improve general health status in participants with long COVID. The study will also seek immune signatures associated with treatment response (overseen by Professor Akiko Iwasaki).

The decentralized study does not require site visits, and participants in all 48 states including the District of Columbia, who meet entry criteria can enroll. It is designed to make it convenient to participate. The study drugs will be delivered to the participant's designated address.

Long COVID is also known as post-acute sequelae of SARS-CoV-2 (PASC).

DETAILED DESCRIPTION:
This decentralized Phase 2, 1:1 randomized, double-blind, superiority, placebo-controlled trial in non-hospitalized symptomatic adult participants with long COVID will investigate the efficacy, safety, and tolerability of 15 days of treatment with nirmatrelvir/ritonavir compared with placebo/ritonavir. The hypothesis is that 15 days of treatment with nirmatrelvir/ritonavir compared with placebo/ritonavir for the treatment of highly symptomatic, adult participants with long COVID will improve their general health as assessed by the National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS)-29 version 2.1 Physical Health Summary Score at Day 28 (2 weeks after the end of the trial drug treatment). This randomized trial is intended to inform future research and will involve an investigation into markers of response.

The primary outcome is the PROMIS-29 Physical Health Summary Score. Secondary outcomes will include the PROMIS subscales and items; the Modified General Symptom Questionnaire (Modified GSQ-30) with PROMIS Cognitive Function v.2.0 - Short Form 6a and supplemental symptoms questionnaire and items; the COVID Core Outcome Measure for Recovery; the EuroQol EQ-5D-5L (USA Version); the Functional Assessment of Chronic Illness Therapy (FACIT)-Item GP5; the Patient Global Impression of Severity (PGIS), Patient Global Impression of Change (PGIC), and symptom assessments and healthcare utilization and death. The trial will also employ immunophenotyping to explore the effects of treatment on immune signatures and immune markers of response. In addition, there will be an evaluation of safety endpoints.

The trial will randomize 100 participants 18 years and older and able to provide legal consent, with long COVID (history of SARS-CoV-2 infection, symptoms consistent with long COVID beginning after the index infection and continuing more than 12 weeks); with a current fair or worse health status and a good or better health status before the index infection and no known other obvious reason for a depressed health status. Exclusion criteria include HIV infection; pregnancy; breastfeeding; renal impairment (eGFR <60 mL/min/1.73 m2); hepatic impairment (Child-Pugh Class B or C); history of clinically significant hypersensitivity reactions [e.g., toxic epidermal necrolysis (TEN) or Stevens-Johnson syndrome] to the product; known or suspected debilitating chronic conditions or those associated with an impaired immune system that pre-date the long COVID syndrome.

ELIGIBILITY:
Inclusion Criteria:

Demographics

* ≥18 years of age and above the age of majority as defined for their state at the time of the screening visit.
* English fluency adequate for communication and able to self-complete the patient-reported outcomes instruments.
* Reside in the 48 contiguous United States

Disease Characteristics

* Prior SARS-CoV-2 infection is required. Documented confirmation of previous COVID-19 infection from either a documented positive PCR test and/or medical records from a healthcare provider (HCP) that coincides with the diagnosis of long-COVID from a healthcare provider.
* Symptoms consistent with long COVID that began within 4 weeks of the index infection and persisted for >12 weeks. These symptoms, according to the World Health Organization definition, 'include fatigue, shortness of breath, cognitive dysfunction but also others, and generally have an impact on everyday functioning. Symptom(s) may be new onset following initial recovery from an acute COVID-19 episode or persist from the initial illness'.
* Baseline "fair" or worse general health status and "good" or better before the index infection and no obvious other reason for the depressed general health status. This is determined from a single-item general health question on the pre-randomization surveys and comorbidity questions.

Surveys and Health Records

• Have connected health records and completed baseline surveys so assessments can be made before randomization of eligibility for the trial. Documentation in the subject's medical record of a physical examination, including vital signs measurement, by a HCP performed after the onset of post-COVID symptoms or within 3 months prior to randomization, whichever is more recent, is required.

Usual Source of Care • Have a usual source of medical care with medical record documentation as required above. (The purpose is to have a health care provider who can be notified of their involvement in the trial and can be a source of care for any adverse effects.)

Informed Consent

• Willing and able to provide informed consent, complete the surveys, clinical assessments, and biospecimen collections. The study does not have sites and participants will not need to travel for any study visits.

Exclusion Criteria Medical Conditions

* HIV infection as determined by laboratory testing at screening.
* Acute medical illness currently or within the past 2 weeks, including COVID-19 infection.
* Known medical history of active liver disease (other than nonalcoholic hepatic steatosis), including chronic or active hepatitis B or C infection, primary biliary cirrhosis, Child-Pugh Class B or C, or acute liver failure. (ALT or ALT level ≥2.5 X ULN or total bilirubin ≥2 X ULN (≥3 X ULN for Gilbert's syndrome) as determined by laboratory testing at screening.
* Receiving dialysis or renal impairment (eGFR estimate <60 mL/min/1.73 m2 ) as determined by laboratory testing at screening.
* Any comorbidity requiring hospitalization and/or surgery within 7 days before trial entry, or that is considered life threatening within 30 days before trial entry, as determined by the Yale team.
* History of hypersensitivity or other contraindication to any of the components of the trial intervention, as determined by the Yale team.
* Other medical or psychiatric condition, in the Yale team's judgment, that makes the participant inappropriate for the trial.
* Immunocompromised, as defined by the CDC; "Examples of medical conditions or treatments that may result in moderate to severe immunocompromise include but are not limited to:

  * Active treatment for solid tumor and hematologic malignancies.
  * Hematologic malignancies associated with poor responses to COVID-19 vaccines regardless of current treatment status (e.g., chronic lymphocytic leukemia, non-Hodgkin lymphoma, multiple myeloma, acute leukemia).
  * Receipt of solid-organ transplant or an islet transplant and taking immunosuppressive therapy.
  * Receipt of chimeric antigen receptor (CAR)-T-cell therapy or hematopoietic stem cell transplant (within 2 years of transplantation or taking immunosuppressive therapy).
  * Moderate or severe primary immunodeficiency (e.g., common variable immunodeficiency disease, severe combined immunodeficiency, DiGeorge syndrome, Wiskott-Aldrich syndrome).
  * Advanced or untreated HIV infection (people with HIV and CD4 cell counts less than 200/mm3, history of an AIDS-defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV).
  * Active treatment with high-dose corticosteroids (i.e., 20 ≥ mg of prednisone or equivalent per day when administered for 2 or more weeks), alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive, tumor necrosis factor blockers, and other biologic agents that are immunosuppressive or immunomodulatory".
* Any concomitant prior chronic condition that has caused debilitating symptoms, even if episodic, such as myalgic encephalomyelitis/chronic fatigue syndrome, chronic Lyme disease, multiple sclerosis, fibromyalgia, mast cell activation disorder, and small fiber neuropathy, postural orthostatic tachycardia syndrome, lupus erythematosus, and others or any prior condition associated with immune dysfunction.

Prior/Concomitant Therapy

* Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance, and for which elevated plasma concentrations may be associated with serious and/or life-threatening events during treatment and for 4 days after the last dose of the trial drugs.
* Concomitant use of any medications or substances that are strong inducers of CYP3A4 are prohibited within 28 days prior to first dose of nirmatrelvir/ritonavir and during trial treatment. A list of these medications will be provided.
* Prior treatment with nirmatrelvir/ritonavir within 2 months prior to randomization.
* Prior treatment with nirmatrelvir/ritonavir at any time if for more than 5 days.
* Individuals who plan to get a COVID-19 vaccine between the time of consent through Day 28 will be excluded from the trial.

Prior/Concurrent Clinical Trial Experience

* Unwillingness to abstain from participating in another interventional clinical study with an investigational compound or device, including those for long COVID therapeutics, through 90 days. (People may be concurrently enrolled in observational studies in general; including the Yale LISTEN study.)
* Previous administration with any investigational drug in a clinical study within 30 days or 5 half-lives preceding the first dose of trial intervention used in this trial (whichever is longer).

Diagnostic Assessments

Known history of any of the following abnormalities within the past 6 months or currently present:

* AST or ALT level ≥2.5 X ULN.
* Total bilirubin ≥2 X ULN (≥3 X ULN for Gilbert's syndrome).
* eGFR <60 mL/min/1.73 m2 within 6 months of the screening visit, using the updated CKD-EPI formula without the race term.
* Absolute neutrophil count <1000/mm3.

Other Exclusions

* Potential participants who are or plan to become pregnant or breastfeeding. Female potential participants will have a pregnancy test during screening.
* Anyone directly involved in the conduct of the trial and their immediate family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS)-29 version 2.1 Physical Health Summary Score | Day 28
  The difference in NIH PROMIS-29 version 2.1 Physical Health Summary Score at Day 28 between nirmatrelvir/ritonavir and placebo/ritonavir treatment estimated with a longitudinal analysis of covariance (ANCOVA) that controls for age, sex, and baseline PROMIS-29 Physical Health Summary Score. PROMIS-29 was selected as a well-validated, non-proprietary general health assessment. PROMIS-29 is a self-report 29-item questionnaire from 7 primary PROMIS domains (depression, physical function, pain interference, fatigue, sleep disturbance, and satisfaction with participation in social roles). PROMIS-29 assessments are transformed into a T-score metric, so that scores have a normal distribution with a population mean T-score of 50 and standard deviation of 10. Higher scores mean better outcomes.

SECONDARY OUTCOMES:
Modified General Symptom Questionnaire-30 (Modified GSQ-30) | Day 28 and at Day 15, and Weeks 6, 10, 14, 18, and 24
  Difference in GSQ-30 between nirmatrelvir/ritonavir and placebo/ritonavir groups. The GSQ-30 is a 30-item questionnaire developed to assess symptom burden over a 2-week time period. The GSQ-30 asks: "how much have you been bothered by any of the following?" with 5 options: "not at all," "a little bit," "somewhat," "quite a bit," and "very much" (scored 0-4); total score ranges from 0 to 120. The GSQ-30 reflects physical and neuropsychiatric symptoms. An additional question (not included in the scoring) asks whether any of the 30 GSQ symptoms have impaired work, social, or family functioning, and asks the rank order of severity (up to 7 items) to identify the symptoms of most concern to the individual. Total score ranges from 0 to 120; a higher score means worse outcome. To align with the other trial questionnaires, we will modified the recall period to 1-week.
PROMIS® Cognitive Function v.2.0 - Short Form 6a | Day 28 and at Day 15, and Weeks 6, 10, 14, 18 and 24
  Difference in PROMIS® Cognitive Function v.2.0 - Short Form 6a between nirmatrelvir/ritonavir and placebo/ritonavir groups. The PROMIS® Cognitive Function v.2.0 - Short Form 6a is a 6-item sub-set scale of the PROMIS® Cognitive Function item bank that assesses patient-perceived cognitive deficits.
COVID Core Outcome Measure for Recovery | Day 28 and at Day 15, and Weeks 14 and 24
  Difference in COVID Core Outcome Measure for Recovery Score between nirmatrelvir/ritonavir and placebo/ritonavir groups. The COVID Core Outcome Measure for Recovery is a single item intended to measure a return to the pre-illness state. Its purpose in this trial is to have a question that directly assesses the participant's perception of their recovery from their SARS-CoV-2 infection. It is scored on a 5-point Likert scale from 0 (completely recovered) to 4 (not recovered at all). Complete recovery means the participant no longer has symptoms related to illness and can do usual daily activities and has returned to their previous state of health and mind (before illness).
EuroQol EQ-5D-5L Utility Score-VAS (USA Version) | Day 28 and at Day 15, and Weeks 14 and 24
  Difference in EuroQol EQ-5D-5L Utility Score and VAS Score between nirmatrelvir/ritonavir and placebo/ritonavir groups. The EQ-5D-5L is a descriptive system in which respondents are asked to report their current state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which has 5 levels of response (no problems, slight problems, moderate problems, severe problems, and extreme problems). There is also a visual analogue scale (VAS). In total there are 6 items. The higher the EQ-VAS score, the better the quality of life.
Functional Assessment of Chronic Illness Therapy (FACIT)-Item GP5 | Day 28 and Day 15
  Difference in FACIT-Item GP5 Score between nirmatrelvir/ritonavir and placebo/ritonavir groups. The single-item FACIT-Item GP5, "I am bothered by side effects of treatment," was included to have a question on the experience with the trial drug and will be prefaced to focus on the trial drug. It is a summary measure of the overall tolerability of treatment, with 5 levels of response: not at all, a little bit, somewhat, quite a bit, and very much. It has a 7-day recall period.
PROMIS-29 Overall and Mental Health Summary Score | Day 28 and at Day 15, and Weeks 6, 10, 14, 18 and 24
  Difference in PROMIS-29 Overall and Mental Health Summary Score between nirmatrelvir/ritonavir and placebo/ritonavir groups. The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and 7 health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using 4 items per domain. There is no total score, but each axis forms its own score. Higher scores mean better outcomes.
Difference in number of hospitalizations and deaths | Day 1 through Week 24 (End of Study)
  Difference in occurrence of hospitalizations and deaths between nirmatrelvir/ritonavir and placebo/ritonavir groups.
Proportion of participants who experience individual Serious Adverse Events (SAE) | up to 6 weeks post starting study drug
  Proportion of participants who experience individual SAEs
Incidence of SAEs leading to discontinuation | Day 15
  The number of SAEs leading to discontinuation in the study
Patient Global Impression of Severity | Baseline, Day 15, Day 28, Week 6, Week 10, Week 14, Week 24
  Based on FDA's recommendations, we will include the Patient Global Impression of Severity (PGIS) and Patient Global Impression of Change (PGIC) scales. These anchor scales can help interpret a clinically meaningful within-patient score change for the key primary and secondary endpoints. We will include two PGIS and two PGIC scales. The PGIS 1 is a single-item questionnaire that asks respondents: "Overall, how would you rate the severity of your long COVID symptoms over the past week?". Responses are: "none," "mild," "moderate," "severe," and "very severe." The PGIS 2 asks "Overall, how would you rate the impact of your symptoms on your overall health over the past week?". Responses are: "none," "mild," "moderate," "severe," and "very severe." The PGISs will be administered at the same intervals as the primary endpoint (PROMIS-29).
Patient Global Impression of Change | Day 15, Day 28, Week 6, Week 10, Week 14, Week 24
  The PGIC 1 asks: "Overall, how would you rate the change in your long COVID symptoms since you started the study?". There 7-point scale options: 1) "very much better", 2) "much better", 3) "minimally better", 4) "no change", 5) "minimally worse", 6) "much worse", or 7) "very much worse". Higher scores indicate a change for the worse. The PGIC 2 asks "Overall, how would you rate your overall health since you started the study?". There 7-point scale options: 1) "very much better", 2) "much better", 3) "minimally better", 4) "no change", 5) "minimally worse", 6) "much worse", or 7) "very much worse". Higher scores indicate a change for the worse. The PGICs will be administered at the same intervals as the primary endpoint (PROMIS-29) with the exception of baseline. These instruments have been used extensively in patient-centered research.

OTHER OUTCOMES:
Exploratory Outcome Measure | Baseline, Day 14 and at Day 28
  Differences in immune signatures between baseline and nirmatrelvir/ritonavir treatment relative to placebo/ritonavir. Immunophenotyping assays will include flow cytometry, multiplex proteomic analysis, linear peptide profiling, and rapid extracellular antigen profiling, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Harlan M Krumholz, MD, SM, Principal Investigator — Yale University; Akiko Iwasaki, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
This plan is pending.

REFERENCES:
- [Derived] Sawano M, Bhattacharjee B, Caraballo C, Khera R, Li SX, Herrin J, Christian D, Coppi A, Warner F, Holub J, Henriquez Y, Johnson MA, Goddard TB, Rocco E, Hummel AC, Mouslmani MA, Hooper WB, Putrino DF, Carr KD, Charnas L, De Jesus M, Nepert D, Abreu P, Ziegler FW 3rd, Spertus JA, Iwasaki A, Krumholz HM. Nirmatrelvir-ritonavir versus placebo-ritonavir in individuals with long COVID in the USA (PAX LC): a double-blind, randomised, placebo-controlled, phase 2, decentralised trial. Lancet Infect Dis. 2025 Aug;25(8):936-946. doi: 10.1016/S1473-3099(25)00073-8. Epub 2025 Apr 3. PMID 40188838